## Assessment of Asthma Management in Children Over 6 Years of Age and Their Caregivers: Implications for the Implementation of the SMART Strategy in Pediatrics

Protocol Version and Date: Version: 1 - Date: 14/05/2025

Protocol Code: IIBSP-EMA-2025-05

Short Title: Asthma Management in Children

Sponsor: Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau – IIB Sant Pau c/

Sant Quintí, 77-79 08041 Barcelona Tel: +34 93 556 56 17 Fax: +34 93 553 78 12

Principal Investigator: Victòria Morón Faura. Pediatric Pulmonology MSc Nurse, Hospital de la Santa Creu i Sant Pau. c/ Sant Antoni Maria Claret, 167. 08025

Barcelona. Tel: +34 647 026 964 E-mail: vmoron@santpau.cat

Confidentiality Statement: This Study Protocol is the property of the Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau – IIB Sant Pau and is a confidential document. It must not be copied or distributed to other parties without prior written authorization from the Institut de Recerca.

## PARTICIPANT INFORMATION SHEET AND INFORMED CONSENT (AGES 11-17)

Study Title: Assessment of Asthma Management in Children Over 6 Years of Age and Their Caregivers: Implications for the Implementation of the SMART Strategy in Pediatrics

Study Code: IIBSP-EMA-2025-05

Principal Investigator: Victòria Morón Faura

Department: Pediatrics Center: Hospital de la Santa Creu i Sant Pau

## PARTICIPANT INFORMATION SHEET

You are invited to participate in this study. This sheet provides information to help you decide whether to participate. Participation is voluntary, and you can withdraw at any time without affecting your medical care.

**Purpose of the Study:** The study aims to determine if a brief educational intervention and nurse demonstration can help you manage your asthma better, use your inhaler correctly, and recognize when it needs to be used.

**Eligibility:** Children aged 6–17 years with a diagnosis of asthma, who have used an inhaler for at least six months, and who attend the Pediatric Pulmonology Clinic at our hospital.

**Study Duration and Visits:** - **Visit 1 (Screening & Baseline):** Eligibility check, basic data collection (age, sex, school), routine breathing tests, inhaler demonstration, simple questionnaires. - **Nurse Education Session:** Practical guidance with illustrated materials on inhaler use, treatment indications, and recognizing worsening asthma. - **Visit 2 (6-Month Follow-Up):** Repeat of previous activities to assess changes.

No additional invasive or painful tests are required beyond standard care.

**Data Protection:** Personal data will be pseudonymized using a code. Only the principal investigator can link the code to your identity. No identifiable information will be disclosed.

**Additional Information:** Data may be used in future related research with your consent. For questions, contact: Mrs. Victòria Morón Faura Pneumoallergy Day Hospital, Floor E, Room B, HSCSP Tel.: 93 291 9000 ext. 8079

| I, (Full Name), have read the information sheet, had the opportunity to ask questions, and received sufficient information about the study. I understand participation is voluntary and may withdraw at any time without affecting my care. | | | |
|---|---|---|---|
| I consent to participate and allow access to my data as described in the information sheet. I authorize the use of collected data in future related studies: $\square$ YES $\square$ NO | | | |
| Participant Signature: Date: | | | ire: |
| PARENT/GUARDIAN INFORMED CONS | | | |
| I, (Parent/Guardian Name), has opportunity to ask questions, and receil understand my child's participation is without affecting care. I freely consent | ave read the infor<br>eived sufficient inf<br>s voluntary and m | mation sheet, had the formation. ay withdraw at any time | _ of |
| I authorize the use of collected data in | future related stu | udies: □ YES □ NO | |
| Parent/Guardian Signature:consents, confirmation that the other pare:Signature: | parent does not o | ppose: Name: | |
| A copy of this form will be kept by both | the participant a | nd the investigator. | |